CLINICAL TRIAL: NCT02624804
Title: A Pilot Study of the Therapeutic Potential of Stem Cell Educator Therapy in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro 6262
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus Type 1
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stem Cell Educator Therapy (Experimental): Patients will have apheresis performed and then have their own blood returned to them with the "educated" lymphocytes
  Interventions: Biological: Stem Cell Educator Therapy

INTERVENTIONS:
Biological: Stem Cell Educator Therapy — Patients will receive apheresis and then have their own blood returned to them with the "educated" lymphocytes
  Other Names: Stem Cell Education

SUMMARY:
This is a prospective, single arm, open-label, single-center pilot study to assess the safety, feasibility, and efficacy of Stem Cell Educator therapy for the treatment of patients with Type 1 Diabetes.

DETAILED DESCRIPTION:
Our previous work demonstrated that human cord blood-derived multipotent stem cells (CB-SCs) are a unique type of stem cell identified from human cord blood, distinct from other stem cell types including hematopoietic stem cells (HSCs), and mesenchymal stem cells (MSCs). The stem cells and harnessed some of their unique properties with Stem Cell Educator therapy by using CB-SCs in a closed-loop system that circulates a patient's blood through a blood cell separator, briefly co-cultures the patient's lymphocytes with adherent CB-SCs in vitro, and returns the "educated" lymphocytes (but not the CB-SCs) to the patient's circulation . This treatment leads to global immune modulations and immune balance as demonstrated by clinical data and animal studies. The Stem Cell Educator therapy may revolutionize the clinical treatment of diabetes and other immune-related diseases through CB-SCs' immune education and induction of immune balance, without the safety and ethical concerns associated with conventional stem cell-based approaches

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years
* Must have a diagnosis of type 1 diabetes mellitus based on the 2015 American Diabetes Association criteria for the Clarification and Diagnosis of diabetes
* Must have a blood test confirming the presence of at least one autoantibody to pancreatic islet cells (IAA, IA2, GAD 65, ZnT8)
* Fasting C-peptide level > 0.3 ng/ml
* Adequate venous access for apheresis
* Ability to provide informed consent
* Must agree to comply with all study requirements and be willing to complete all study visits

Exclusion Criteria:

* AST or ALT 2 > x upper limit of normal.
* Creatinine > 2.0 mg/dl.
* Known coronary artery disease or EKG suggestive of coronary artery disease unless cardiac clearance for apheresis is obtained from a cardiologist.
* Known active infection
* Pregnancy or breastfeeding mothers
* Use of immunosuppressive medication within one month of enrollment including but not limited to prednisone, cyclosporine, tacrolimus, sirolimus, and chemotherapy.
* Presence of any other autoimmune diseases (lupus, rheumatoid arthritis, scleroderma, etc.)
* Anticoagulation other than ASA.
* Hemoglobin < 10 g/dl or platelets < 100 k/ml
* Is unable or unwilling to provide informed consent
* Presence of any other physical or psychological medical condition that, in the opinion of the investigator, would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Donato, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Educator Therapy
Started | 13
Completed | 8
Not Completed | 5
Not completed — Screen Failure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Stem Cell Educator Therapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 24 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events
Description: The primary study endpoint will be the occurrence of treatment-related adverse effects. Adverse events that occur during therapy (especially those that necessitate temporary or permanent discontinuation of therapy) and over the 12-month follow-up period will be assessed.
Time Frame: 12 months
Population: Patients Experiencing Treatment Related Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Educator Therapy
Number analyzed (Participants) | 8
Participants | 1

2. Secondary Outcome: Number of Patients Unable to Complete Therapy
Description: Number of patients who were unable to complete SCE Therapy.
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Educator Therapy
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: From the initiation of any study procedures to the end of the study treatment follow-up, up to 24 months.
Arm/Group | Stem Cell Educator Therapy
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Educator Therapy (N=8)
Depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Educator Therapy (N=8)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Body Aches (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Infection Strep Throat (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT02624804/Prot_SAP_000.pdf